CLINICAL TRIAL: NCT01428388
Title: Comparison of Anti-vascular Endothelial Growth Factors Agents in the Treatment of Macular Edema Following Retinal Vein Occlusion
Brief Title: Bevacizumab Versus Ranibizumab in Treatment of Macular Edema From Vein Occlusion
Acronym: CRAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barnes Retina Institute (Other)
Collaborators: Retina Associates of Florida, P.A. (Other); Illinois Retina Associates (Other); Kresge Eye Institute (Other); Long Island Vitreoretinal Consultants (Other); Mid Atlantic Retina (Other); Retina Associates, Kansas City (Other); Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Rhonda Weeks, Gaurav Shah, MD, Barnes Retina Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRAVE1
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Retinal Vein Occlusion; Macular Edema
Keywords: macular edema; vein occlusion; bevacizumab; ranibizumab; vascular endothelial growth factor
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab (Active Comparator)
  Interventions: Drug: Intravitreal injection of bevacizumab
- Ranibizumab (Active Comparator)
  Interventions: Drug: Intravitreal injection of ranibizumab (0.5 mg per dose)

INTERVENTIONS:
Drug: Intravitreal injection of bevacizumab — 1.25 mg per dose, delivered monthly by intravitreal injection for six months
  Arms: Bevacizumab
Drug: Intravitreal injection of ranibizumab (0.5 mg per dose) — 0.5 mg per dose, delivered monthly by intravitreal injection for six months
  Arms: Ranibizumab

SUMMARY:
Antagonists of the vascular endothelial growth factor (VEGF) pathway are effective in treating macular edema resulting from retinal vein occlusion (RVO). In the eye, the two most widely used anti-VEGF agents are ranibizumab and bevacizumab. Only ranibizumab has been FDA-approved for the treatment of macular edema from RVO, however bevacizumab has been used off-label by many ophthalmologists with good success. Furthermore, the cost of bevacizumab is less than one-tenth the cost of ranibizumab. Here the investigators conduct a six month randomized, prospective interventional trial comparing the effectiveness of ranibizumab with bevacizumab in the treatment of macular edema from RVO. Primary outcome measures are change in central retinal thickness. Secondary measures are change in visual acuity from baseline and change in angiographic properties of macular lesions from baseline after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Visual acuity of 20/40 - 20/320 in the study eye (regardless of relative APD)
* Central foveal thickness (CFT) of > 250 microns as assessed by OCT (see below)
* Diagnosis of retinal vein occlusion in the past 9 months
* Age over 50 years

Exclusion Criteria:

* History of previous intraocular surgery in the study eye, including pars plana vitrectomy (but not including uncomplicated cataract surgery), within 60 days of the screening visit
* Inability to make study visits
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure (IOP) ≥ 25 mmHg) despite treatment with two or more topical pharmacological anti-glaucomatous medication)
* Pregnancy or lactation
* Evidence of any diabetic retinopathy on exam or history of diabetic macular edema within 12 weeks of study onset
* Any intravitreal injections within 12 weeks of study onset
* Prior retinal vein occlusion
* History of pan-retinal photocoagulation within 3 months of study onset or anticipated within 4 months after study onset
* History of cerebrovascular event or myocardial infarction within 3 months of study onset

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
change in central retinal thickness | six months compared to baseline
  central thickness is measured using optical coherence tomography (OCT)

SECONDARY OUTCOMES:
change in best-corrected Snellen visual acuity | six months compared to baseline
  best-corrected Snellen visual acuity (BCVA) is the best visual acuity measured using a standard Snellen eye chart at 20 feet between (1) uncorrected vision, (2) vision with current eyeglasses or (3) pinholed visual acuity.
change in fluorescein angiogram | six months compared to baseline
  fluorescein angiograms will measure area of peripheral nonperfusion. This will be interpreted by a designated physician at each testing center.

CONTACTS AND LOCATIONS:
Locations (1):
- The Retina Institute, St Louis, Missouri, United States

REFERENCES:
- [Derived] Rajagopal R, Shah GK, Blinder KJ, Altaweel M, Eliott D, Wee R, Cooper B, Walia H, Smith BT, Joseph DP. Bevacizumab Versus Ranibizumab in the Treatment of Macular Edema Due to Retinal Vein Occlusion: 6-Month Results of the CRAVE Study. Ophthalmic Surg Lasers Imaging Retina. 2015 Sep;46(8):844-50. doi: 10.3928/23258160-20150909-09. PMID 26431300